CLINICAL TRIAL: NCT05154474
Title: Assessment of the Proportion of Patients With Sarcopenia at Diagnosis for Patients With Previously Untreated Metastatic Cancer or Hematologic Malignancy.
Brief Title: Assessment of Sarcopenia at Diagnosis for Patients With Previously Untreated Metastatic Cancer or Hematologic Malignancy
Acronym: SPACE2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Weprom (Other)
Responsible Party: Sponsor
Other Study IDs: WP-2021-03; 2021-A01670-41 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2021-11-29; First posted 2021-12-13 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Cancer; Cancer, Breast; Cancer Colon; Cancer, Rectum; Cancer, Lung; Cancer Ovaries; Cancer Prostate; Cancer, Kidney; Cancer Pancreas; Myeloma; Myelodysplasia; Leukemia, Myeloid, Acute; Leukemia,Myeloid, Chronic; Leukemia, Lymphocytic, Acute; Leukemia, Lymphocytic, Chronic
Keywords: sarcopenia; quality of life questionnaire; nutrition
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Kidney Neoplasms; Pancreatic Neoplasms; Neoplasms, Plasma Cell; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard: Standard follow-up MNA, IPAQ, SARC-F and SarQOL questionnaire
  Interventions: Other: Standard

INTERVENTIONS:
Other: Standard — Standard follow-up with clinical exams, functionnal test at baseline, Ct scan MNA, IPAQ, SARC-F and SarQOL questionnaires

SUMMARY:
Sarcopenia is defined as reduction in muscle mass and function according to the criteria of the European Working Group on Sarcopenia in older people. Initially described for elderly patients, it is also presented as a negative prognostic factor in overall survival in oncology in certain locations (lung, ENT pathways, colon, pancreas) and more controversially for hemopathies. Its screening by measurement of skeletal muscle mass by CT scan and / or PET scan against L3 and by physical functional tests is not routinely integrated despite international recommendations. Sarcopenia is one of the characteristics of patient fragility that can induce more complications, lengthen the average length of hospital stay and reduce overall survival. The PRONOPALL score, a predictor score for survival validated by a previous study, will be correlated with the presence (or absence) of sarcopenia at inclusion for patients with a solid tumor (breast, ovary, prostate cancer , kidney, lungs, pancreas, colorectal). A prospective study on 38 patients with metastatic cancer was carried out at the Victor Hugo clinic in Le Mans between 01/JUN/21 and 31/AUG/21 (SPACE, ClinicalTrials.gov number, NCT04714203): 25 patients were analyzable on the CT and PRONOPALL score data with a prevalence of sarcopenia of 60% and median overall survival of 14 months (unpublished data), clinical performance and muscle strength tests were not carried out (as in the publications cited above).

A prospective study for the detection of sarcopenia is indicated by extending to blood diseases with the integration of clinical tests included in the initial APA (Adapted physical activity) assessment recommended for diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years or older
2. Patient with solid cancer diagnosed with metastatic disease,or hematological disease requiring treatment (myeloma, lymphoma, high-risk myelodysplasia, acute or chronic myeloid leukemia, acute and chronic lymphoid leukemia)
3. Patient naive of cancer treatment
4. Pathology including performing a CT scan with cuts of the lumbar spine in standard care
5. Patient enrolled in social security
6. Patient has given his written consent ahead of any specific protocol procedure.

Exclusion Criteria:

1. Minor patient
2. Metastatic neurological impairment
3. Patient deprived of their liberty, under guardianship or trusteeship
4. Patient with dementia, mental disorders or psychological pathology which could compromise patient informed consent and/or the observance of the study protocol
5. Patient cannot submit to the protocol for psychological, social, familial or geographical reasons
6. Patient is pregnant
7. History of cancer treated (excluding surgery alone for tumors in situ) within 5 years of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited during medical consultations or hospitalization in an onco-hematology service
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with sarcopenia diagnosed with metastatic cancer. | At inclusion
  Sarcopenia is defined for those under 60 years of age by LMSI<43.1 cm²/m² for men and <32.7 cm²/m² for women, and for patients over 60 years of age by <38.6 cm²/m² for men and <30.7 cm²/m² for women..

SECONDARY OUTCOMES:
Overall Survival | 18 months
  Calculated from the date of inclusion to the date of death due to any cause or the date last known to be alive if patient is censored.
Event Free survival | 18 months
  Calculated from the date of start of treatment to the date of first event (progression, death, infectious complications, thrombosis, side effects of treatments of grade 2 or higher)
Progression Free survival | 18 months
  Calculated from the date of start of treatment to the date of first progression of disease based on Investigator assessment or the date of death or censored at the date of the last valid tumor assessment before start of a new therapy for patients who are still alive and without progression
Unanticipated hospitalization rate | 18 months
  Calculated from the date of start of treatment for all unplanned hospitalizations for side effects of treatments of grade 2 or higher, infectious complications, thrombosis, relapse or progression
Statistical relationship between sarcopenia and the PRONOPALL score | 18 months
  For the cancer subtypes concerned (breast, colon, rectum, lungs, ovaries, prostate, kidney, pancreas)
Rate of undernourished patients | 18 months
  Calculated according to WHO classification
Rate of patients with sarcopenia at diagnosis across the inclusive population | 18 months
  Calculated from the number of patients who were screened for sarcopenia at diagnosis in the active file of patients meeting the inclusion criteria in all participating centers

CONTACTS AND LOCATIONS:
Overall Officials: Katell LE DU, MD, Principal Investigator — Private Hospital of Confuent, Nantes
Locations (2):
- France (2):
  - Clinique Victor Hugo/Centre Jean Bernard, Le Mans
  - Clinique privé du Confluent, Nantes

IPD SHARING:
Plan to Share IPD: No